CLINICAL TRIAL: NCT03585413
Title: Impact of a Specific Micronutrient-probiotic-combination on Fatty Liver and Cardiometabolic Status of Obese Patients After Mini-Gastric Bypass Surgery
Brief Title: Impact of a Specific Micronutrient-probiotic-supplement on Fatty Liver of Patients After Mini-Gastric Bypass Surgery
Acronym: FMG-01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bonn Education Association for Dietetics r.A., Cologne, Germany (Industry)
Collaborators: St. Franziskus Hospital (Other); University of Bonn (Other); FormMed HealthCare AG (Unknown)
Responsible Party: Principal Investigator, Karl Peter Rheinwalt, Scientific Adviser for Visceral- and Metabolic Surgery, Bonn Education Association for Dietetics r.A., Cologne, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BFD-02/FMG-01
Record Dates: First submitted 2018-06-07; First posted 2018-07-13 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Obesity; Gastric Bypass; NAFLD
Keywords: Bariatric surgery; Obesity; NAFLD; Micronutrient supplementation; Probiotic supplementation
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: prospective, randomized, placebo-controlled, double-blind interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific Micronutrient-probiotic-combination (Active Comparator): Intake of one micronutrient capsule three times daily and probiotic powder twice daily starting on the first day after hospital discharge until 12 weeks postoperatively.
  The micronutrient capsules consist of vitamins, minerals, phytochemicals and bioactive substances. The probiotic supplement is a powder of 10 different species of probiotic bacteria.
  Interventions: Dietary Supplement: Micronutrient-probiotic-combination
- Micronutrient-placebo-combination (Placebo Comparator): Intake of one micronutrient capsule three times daily and placebo powder twice daily starting on the first day after hospital discharge until 12 weeks postoperatively.
  The micronutrient-control-combination consists of a micronutrient capsule (vitamins and minerals) but without phytochemicals and bioactive substances, and a placebo powder manufactured to mimic the probiotic powder.
  Interventions: Dietary Supplement: Micronutrient-placebo-combination

INTERVENTIONS:
Dietary Supplement: Micronutrient-probiotic-combination — Specific combined micronutrient-probiotic-supplement with different vitamins, minerals, phytochemicals and bioactive substances, and a mixture of 10 different probiotic bacteria.
  Arms: Specific Micronutrient-probiotic-combination
Dietary Supplement: Micronutrient-placebo-combination — micronutrient (capsule)-placebo (powder)-supplement
  Arms: Micronutrient-placebo-combination

SUMMARY:
Aim of this prospective randomized intervention study is to evaluate the effect of a dietary intervention with a specific micronutrient-probiotic-combination for 12 weeks on fatty liver and cardiometabolic status in obese, nonalcoholic fatty liver disease (NAFLD) patients after Mini-Gastric Bypass (MGB) surgery.

DETAILED DESCRIPTION:
Background:

The increasing prevalence of obesity and diabetes mellitus seems to reach epidemic proportions worldwide. In particular visceral obesity in combination with impaired glucose tolerance is associated with risk for progression of a broad spectrum of cardiometabolic diseases such as type 2 diabetes, hypertension, dyslipidemia, cardiovascular disease and non-alcoholic fatty liver disease (NAFLD). Thus, among patients undergoing bariatric surgery more than 95% have NAFLD, with nonalcoholic steatohepatitis (NASH) being present in 32-39 %.

Only bariatric surgery currently seems to attain long-term weight loss in morbidly obese patients. In addition, greater success in terms of improvement in obesity related comorbidities and reduction of overall-mortality can be achieved by surgical measures. Recent data indicate that Mini-Gastric Bypass (MGB) is an effective procedure for weight loss and reduction of comorbidities. Although weight loss is usually recommended as therapy for obesity with NAFLD and NASH, not all NAFLD patients benefit from surgical induced weight loss as indicated by increase in transaminase activity. An optimized micronutrient in combination with a probiotic supplementation could be a useful tool to prevent the transition from NAFLD to NASH.

Aim:

Therefore this study aims to elucidate the effect of a specific micronutrient-probiotic-combination on fatty liver and insulin resistance in obese patients after MGB surgery. Furthermore, this study aims to help optimizing the dietary food supplementation after MGB to reduce the progress of NAFLD/NASH and cardiometabolic diseases.

Methods:

A randomized double blind clinical trial of 12 week dietary intervention with a specific micronutrient-probiotic-combination will be conducted in obese patients with NAFLD after standardized MGB surgery. To this end, a total of 60 patients will be randomly assigned to a specific micronutrient-probiotic-combination or micronutrient-placebo-combination group. During the preoperative 4-week run-in phase, each patient receives a formula diet to improve protein and micronutrient supply. This should align the metabolic situation within the study group. At baseline and study end blood samples are taken for further analysis of metabolic, clinical and biochemical parameters. Anthropometric data (body height, body weight, and waist circumference) and bioelectrical impedance analysis are also collected at the beginning and after 8 and 12 weeks. Fecal samples will be collected prior to surgery and after 4, 8 and 12 weeks (concomitant variable). All patients will fill out validated food intake questionnaires and stool questionnaires (frequency and consistence) after 4, 8 and 12 weeks (concomitant variable).

ELIGIBILITY:
Inclusion Criteria:

* subjects 20-65 years old
* BMI ≥ 35 kg/m² to ≤ 50 kg/m²
* Fatty Liver Index ≥ 60

Exclusion Criteria:

* subjects with anamnestic known alcoholic-fatty liver disease, hepatitis B, hepatitis C, HIV/ AIDS
* subjects with chronic conditions such as active malignant disease, inflammatory bowel disease and other systemic inflammatory conditions
* supplementation with dietary supplements or drugs which contain probiotics, milk thistle, fatty acids, vitamins or minerals 4 weeks before bariatric surgery
* treatment with psychotropic drugs
* diabetic patients who are treated with antidiabetic medications
* use of antibiotic 4 weeks before bariatric surgery
* weight gain during run-in phase of more than 5 %
* in women of childbearing age, pregnancy or breastfeeding
* no safe method of contraception in women of childbearing age

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Change in alanine-aminotransferase (ALAT) activity in serum | Baseline and 12 weeks
  ALAT in U/l

SECONDARY OUTCOMES:
Change in Fatty Liver Index (FLI) | Baseline and 12 weeks
  FLI will be calculated as: [e 0.953 x loge (triglycerides (mg/dl)) + 0.139 x BMI (kg/m²) + 0.718 x loge (GGT (U/l)) + 0.053 x waist circumference (cm) - 15.745) / (1 + e 0.953 x loge (triglycerides (mg/dl)) + 0.139 x BMI (kg/m²) + 0.718 x loge (GGT (U/l)) + 0.053 x waist circumference (cm) - 15.745)] × 100.
  A FLI < 30 rules out fatty liver and a FLI > 60 rules in fatty liver.
Change in nonalcoholic fatty liver disease (NAFLD) Fibrosis Score (NFS) | Baseline and 12 weeks
  NFS will be calculated as: - 1.675 + 0.037 x age (years) + 0.094 x BMI (kg/m²) + 1.13 x impaired fasting glucose (IFG)/diabetes (yes = 1, no = 0) + 0.99 x aspartate aminotransferase (ASAT)/ALAT ratio - 0.013 x platelet (x10^9) - 0.66 x albumin (g/dl).
  NFS > 0.676 is considered to be diagnostic for the presence of significant fibrosis.
  NFS < -1.455 is considered to be diagnostic fot the absence if fibrosis. NFS scores between -1.455 and 0.675 are referred as "indeterminate" scores.
Change in fasting glucose concentration | Baseline and 12 weeks
  Fasting glucose in mmol/l
Change in fasting insulin concentration | Baseline and 12 weeks
  Fasting insulin in pmol/l
Change in homeostatic model assessment (HOMA) of insulin resistance (IR) (HOMA-IR) | Baseline and 12 weeks
  HOMA-IR will be calculated as: fasting insulin (μU/ml) x fasting glucose (mmol/l) / 22.5.
  HOMA-IR > 2.77 is considered to be diagnostic for insulin resistance.
Change in glycated haemoglobin (HbA1c) | Baseline and 12 weeks
  Intervention change in HbA1c level
Change in resting blood pressure | Baseline and 12 weeks
  Intervention changes in resting blood pressure in mmHg
Change in heart rate | Baseline and 12 weeks
  Intervention changes in heart rate in bpm

CONTACTS AND LOCATIONS:
Overall Officials: Karl Peter Rheinwalt, MD, Principal Investigator — St. Franziskus Hospital, Cologne and Bonn Education Association for Dietetics r.A., Cologne, Germany
Locations (1):
- St. Franziskus-Hospital, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crommen S, Rheinwalt KP, Plamper A, Rosler D, Weinhold L, Metzner C, Egert S. Prognostic Characteristics of Metabolic Dysfunction-Associated Steatotic Liver in Patients with Obesity Who Undergo One Anastomosis Gastric Bypass Surgery: A Secondary Analysis of Randomized Controlled Trial Data. Nutrients. 2024 Sep 23;16(18):3210. doi: 10.3390/nu16183210. PMID 39339810
- [Derived] Crommen S, Rheinwalt KP, Plamper A, Simon MC, Rosler D, Fimmers R, Egert S, Metzner C. A Specifically Tailored Multistrain Probiotic and Micronutrient Mixture Affects Nonalcoholic Fatty Liver Disease-Related Markers in Patients with Obesity after Mini Gastric Bypass Surgery. J Nutr. 2022 Feb 8;152(2):408-418. doi: 10.1093/jn/nxab392. PMID 34919684